CLINICAL TRIAL: NCT00735150
Title: Awareness and Attitudes Regarding Prenatal and Preimplantation Genetic Diagnosis for Inherited Breast/Ovarian Cancer Risk
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The New School for Social Research (Other); Hadassah Medical Organization (Other); New York University (Other); New York Presbyterian Hospital (Other)
Responsible Party: Karen Hurley, PhD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 06-137
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Breast; Ovary; Mutation carrier
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: 25 female and 5 male BRCA carriers
  Interventions: Behavioral: questionnaire, interview

INTERVENTIONS:
Behavioral: questionnaire, interview — You will be asked to make a one-time visit to MSKCC. At that research visit, you will be asked to complete a short questionnaire about your knowledge of various reproductive technologies relevant to individuals at hereditary risk. Then you will watch a short presentation about these reproductive technologies and complete a second brief questionnaire to assess your understanding of the presentation. Afterwards, you will meet with an interviewer one-on-one for about one hour, during which time you may share your thoughts and feelings about the use of these reproductive technologies.

SUMMARY:
We are inviting you to participate in a study of how people who have had genetic counseling for breast/ovarian cancer risk feel about certain reproductive technologies, preimplantation genetic diagnosis (PGD) and prenatal genetic diagnosis (PND), that may reduce the chances of passing increased risk onto one's children. We would also like feedback from patients who have been to our clinic in the past on the best ways to talk about PGD and PND during genetic counseling sessions. We are seeking both the opinions of people who are interested in these technologies and those who are not. It does not matter whether you have heard of PGD or PND before - you can still participate. Your past experience with genetic counseling is valuable to us in deciding how to communicate this information during sessions.

ELIGIBILITY:
Inclusion Criteria:

* Females and males who are carriers of deleterious mutations in the genes BRCA1 or BRCA2.
* Over age 18 and:

  1. For women, less than 43
  2. For men, less than 50.
* Received genetic testing and counseling for BRCA.
* Fluent in English.

Exclusion Criteria:

* Patients who are currently under treatment (chemotherapy, radiation)
* Individuals who refuse to discuss reproductive issues.
* Unable to give informed consent due to physical, cognitive, or psychiatric disability

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Prospective participants will be recruited through the MSKCC clinics that serve high-risk patients (e.g. Clinical Genetics Service, Special Surveillance Breast Program, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To explore the attitudes of BRCA1/2 mutation carriers about PGD/PND, most notably benefits and drawbacks, as well as ethical and emotional considerations; | conclusion of study

SECONDARY OUTCOMES:
To elicit opinions from patients who have previously undergone BRCA1/2 genetic counseling as to when and how information about PGD/PND should be presented (e.g., timing, level of detail,etc) | conclusion of study
To explore whether different themes emerge for subgroups of patients (completed childbearing vs. not; affected vs. unaffected). | conclusion of study
To gain preliminary data on themes that might be particularly important to male BRCA1/2 carriers. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hurley, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org